CLINICAL TRIAL: NCT05640713
Title: A Single Dose-escalation Study to Evaluate the Safety and Efficacy of Allogeneic CAR-T Targeting CD19 (ThisCART19A) in Adult Patients With B Cell Malignancies After Failure of Autologous Chimeric Antigen Receptor T- Cell(CAR-T) Therapy
Brief Title: Assessment of Safety and Efficacy of ThisCART19A in Adult Patients With B Cell Malignancies After Failure of Autologous Chimeric Antigen Receptor T- Cell(CAR-T) Therapy
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Collaborators: Fundamenta Therapeutics, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ThisCART19A （FT400-011）
Record Dates: First submitted 2022-11-28; First posted 2022-12-07 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-11

CONDITIONS: Allogeneic, CAR-T, Protein Sequestration, Non-gene Edited
MeSH Terms: interventions — fludarabine; Cyclophosphamide; CBV protocol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ThisCART19A cells infusion (Experimental): In this study, allogeneic anti-CD19 CAR T cell (ThisCART19A) infusion is used to treat patients with refractory or relapsed CD19 positive B cell acute lymphoblastic leukemia.
  Interventions: Drug: ThisCART19A; Drug: Fludarabine Pill; Drug: Cyclophosphamide; Drug: VP-16 Protocol

INTERVENTIONS:
Drug: ThisCART19A — ThisCART19A is a new type CAR-T therapy for patients with r/r B Cell Malignancy .
Drug: Fludarabine Pill — Fludarabine is used for lymphodepletion.
Drug: Cyclophosphamide — Cyclophosphamide is used for lymphodepletion.
Drug: VP-16 Protocol — VP-16 is used for lymphodepletion.

SUMMARY:
This is a a phase 1, open label study to assess the safety and efficacy of ThisCART19 (Allogeneic CAR-T targeting CD19) in adult patients with B cell malignancies after failure of autologous chimeric antigen receptor T- cell(CAR-T) therapy in china.

DETAILED DESCRIPTION:
This is a phase 1, single-center, nonrandomized, open-label, dose-escalation and dose expansion study to evaluate the safety and efficacy of ThisCART19A in adult patients with B cell malignancies after failure of autologous chimeric antigen receptor T- cell(CAR-T) therapy and identify a treatment regimen most likely to result in clinical efficacy while maintaining a favorable safety profile.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with relapsed or refractory acute lymphocytic leukemia, or lymphoma；
2. No gender limitation, Age 14 years to 75 years (both upper and lower limits included)；
3. Failing to autologous CAR-T therapy；
4. Should be confirmed Cluster of differentiation(CD)19 positive；
5. The expected survival time is ≥12 weeks;
6. ECOG score 0-1;
7. Measurable or detectble disease at time of enrollment.
8. Adequate bone marrow, renal, hepatic, pulmonary and cardiac function；

Exclusion Criteria:

1. Allergic to preconditioning measures；
2. Patients with other malignancies other than B-cell malignancies within 5 years prior to screening. Patients with cured skin squamous carcinoma, basal carcinoma, non-primary invasive bladder cancer, localized low-risk prostate cancer, in situ cervical/breast cancer can be recruited；
3. Uncontrollable bacterial, fungal and viral infection during screening；
4. Patients had pulmonary embolism (PE) and/or deep vein thrombosis (DVT) within 3 months prior to enrollment;
5. Had intolerant severe cardiovascular and cerebrovascular diseases and hereditary diseases prior to enrollment；
6. The presence of central nervous system involvement；
7. Active hepatitis B virus (HBV) or hepatitis C virus (HCV) or Human immunodeficiency virus (HIV) or Syphilis infection. HBV-DNA < 2000 IU/mL can be enrolled, but should admitted to use anti-virus drugs such as entecavir, tenofovir, etc, and supervisory the relative indication during the treatment；
8. Had big lesion(single lesion diameter ≥10 cm)；
9. Receive allogeneic hematopoietic stem cell transplantation less than 100 days；
10. Vaccinated with influenza vaccine within 2 weeks prior to cleansing (SARS-COV19 can be included, inactivated, live/non-live adjuvant vaccinations allowed to be included)；
11. Patients who are receiving GvHD treatment; Patients without GvHD and who had stopped immunosuppressive drugs for at least 1 month were eligible for inclusion；
12. Women who are in pregnant or lactating, and female subjects or partners who plan to be pregnant within 1 year after cell infusion. Male subjects who plan pregnancy within 1 year after infusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Dose limited toxicity(DLT) observation in patient with B Cell Malignancy in each dose level during dose escalation stage | 28 days
  DLT is defined as the incidence of severe adverse events related to ThisCART19A more than 33% in each dose level.
Objective Response Rate within 3 months during dose expansion stage | 3 months
  For Acute Lymphoblastic Leukemia (ALL), Objective response rate(ORR) is the percentage of patients who achieve Complete Response (CR) or Complete Response With Incomplete Hematologic Recovery (CRi); for lymphoma, ORR is the incidence of either a complete response (CR) or a partial response (PR).
Minimum Residual Disease (MRD) Negative Remission Rate within 3 months during dose expansion stage | 3 months
  MRD was assessed utilizing multicolor flow cytometry to detect residual cancerous cells with a sensitivity of 10^-4. MRD negative remission was defined as MRD < 10^-4 threshold. Percentage of participants with MRD negative remission was reported.

SECONDARY OUTCOMES:
Duration of response(DOR) during dose escalation stage and expansion stage | 24 months
  DOR was defined as the time from first CR/CRi or PR to relapse or any death in the absence of documented relapse.
Relapse-free Survival (RFS) | 24 months
  RFS is defined as the time from the date of ThisCART19A infusion to the date of disease relapse or death from any cause.
Event-free Survival (EFS) | 24 months
  EFS is defined as the time from the date of ThisCART19A infusion to the date of disease relapse, progression, genetic relapse or death from any cause.
Overall Survival (OS) | 24 months
  OS is defined as the time from the date of ThisCART19A infusion to the date of death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Henan cancer hospital, Zhengzhou, Henan, China